CLINICAL TRIAL: NCT06114615
Title: Digital Monitoring for Patients Post Coronary Interventions to Reduce Risk for Recurrent Adverse Cardiovascular Events
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1972752
Record Dates: First submitted 2023-10-12; First posted 2023-11-02 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
Keywords: post-PCI; digital monitoring; cardiac rehabilitation
MeSH Terms: conditions — Coronary Artery Disease | interventions — Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Discharged with LiveCare and Text Message Intervention (Active Comparator): Patients receive blood pressure monitoring and text messages reminders for enrollment in cardiac rehab, follow up appointment, diet and exercise counseling.
  Interventions: Device: LiveCare; Behavioral: Text Messages
- Discharged with Conventional Care (Sham Comparator): Patients do not receive blood pressure monitoring and text messages reminders for enrollment in cardiac rehab, follow up appointment, diet and exercise counseling.
  Interventions: Other: Conventional Care

INTERVENTIONS:
Device: LiveCare — Patient use LiveCare device to monitor their blood pressure and data is transmitted to dashboard.
  Other Names: Blood Pressure and Weight Monitoring
  Arms: Discharged with LiveCare and Text Message Intervention
Behavioral: Text Messages — Patients also receive text messages after their PCI procedure for follow up appointment reminders, enrollment in cardiac rehab, and diet and exercise counseling.
  Arms: Discharged with LiveCare and Text Message Intervention
Other: Conventional Care — No digital monitoring with LiveCare device and no text messages.
  Arms: Discharged with Conventional Care

SUMMARY:
The study aims to support patients immediately after percutaneous coronary intervention (PCI) by implementing a telemonitoring program. Eligible patients have coronary heart disease and undergo PCI. The intervention group receives remote monitoring and text-based follow-up, with established health goals and education on using the telemonitoring application, along with necessary devices. The control group gets standard care. Outcomes measured include blood pressure, LDL levels, patient satisfaction, revascularization, and mortality. The study findings will enhance patient care after PCI and contribute evidence for widespread telemonitoring implementation in healthcare systems, aiding medical therapy and lifestyle modifications.

DETAILED DESCRIPTION:
The study involves 200 participants divided into intervention and control groups, all diagnosed with coronary heart disease and treated with PCI. Upon discharge, the intervention group receives remote monitoring, text messages, and devices for self-management. Control group receives standard care. Recruitment is from cardiology and primary care clinics, with interpreters available. Study coordinator guides device setup during enrollment. Intervention group receives daily messages for a week, then weekly reminders and counseling. Messages are in English or Spanish as per preference. Patient data is collected, including demographics, medications, and outcomes such as blood pressure and readmission rates. Satisfaction is evaluated through surveys and interviews.

ELIGIBILITY:
Inclusion Criteria:

* Includes patients with coronary heart disease diagnosis and treatment with PCI who follow up at University of California Davis Health.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
blood pressure, systolic and diastolic | 1 month, 6 months
readmission rate | 1 month, 6 months
enrollment rate in cardiac rehabilitation | 1 month, 6 months
rate of non-compliance to medications prescribed at discharge | 1 month, 6 months
average ratings on the telehealth usability questionnaire | six months
  assess patient satisfaction with the teleheath program with 12 questions, each 1-7 points. Total of 84 points; higher score indicates greater satisfaction
patient rate of first follow up appointment | 1 month, 6 month

SECONDARY OUTCOMES:
lipid profile | one month, six months
Major adverse cardiovascular events (MACE) | one month, six months

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis Medical Center Division of Cardiovascular Medicine, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No